CLINICAL TRIAL: NCT05814003
Title: The Clinical Effectiveness of Hydroxylated Polymethoxy Flavones Solid Dispersion as a Dressing Material for Palatal Graft Donor Sites
Brief Title: Clinical Effectiveness of Polymethoxy Flavones Solid Dispersion as a Dressing Material for Palatal Grafts Donor Sites
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mortada, associate professor - faculty of dentistry, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HW37
Record Dates: First submitted 2022-10-10; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Soft Tissue Infections; Gingival Recession
MeSH Terms: conditions — Soft Tissue Infections; Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hydroxylate flavones (Experimental): flavonoids mainly derived from citrus peel and have numerous strong biological activities, including anti-inflammatory , antioxidant , antimicrobial , and anticancer
  Interventions: Drug: hydroxylate flavones solid dispersion application; Other: Placebo
- alveogyl (Active Comparator): ALVOGYL is a brown fibrous paste which contains per 100 g the following active ingredients : 25.70 g of butamben, 15.80 g of iodoform and 13.70 g of eugenol.
  Interventions: Drug: hydroxylate flavones solid dispersion application; Other: Placebo
- stent (Placebo Comparator): acrylic resin material used to cover denuded soft tissues
  Interventions: Drug: hydroxylate flavones solid dispersion application

INTERVENTIONS:
Drug: hydroxylate flavones solid dispersion application — this drug has the antibacterial and anti inflammatory actions could help the palatal donor sites to promote the wound healing
  Other Names: Natural therapy without side effects
Other: Placebo — Dough inert material without any therapeutic action
  Arms: alveogyl; hydroxylate flavones

SUMMARY:
Free gingival grafting surgeries require palatal grafts harvesting from the patient own palates . The donor sites pain , infection and retarded healing by secondary intension are the complication .

DETAILED DESCRIPTION:
After the preparation and characterization of the solid dispersion of hydroxylated methoxy flavones, free gingival grafting surgeries require palatal grafts harvesting from the patient own palates . The donor sites pain , infection and retarded healing by secondary intension are the complications ; the aim of the study is to assess the analgesic , anti inflammatory effects of hydroxylated methoxy flavones.

ELIGIBILITY:
Inclusion Criteria:

* insufficient zone of keratinized gingiva recession of the gingiva non smokers free from systemic disorders

Exclusion Criteria:

* smokers insufficient palatal donor sits un realistic expectations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
post operative pain (VAS scale) | first day postoperative to 30 days (days)
  VAS scale from 0 no pain to 10 excruciating pain (healing)

SECONDARY OUTCOMES:
Number of analgesic and anti inflammatory pills consumed | first day postoperative to 30 days (days)
  Minimizing the pain and inflammation during healing process post operative swelling

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mortada, Professor, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paolantonio M, De Ninis P, Secondi L, Femminella B. The Full-Thickness Palatal Graft Technique: Description of an Original Surgical Technique and 15 Case Reports. Int J Periodontics Restorative Dent. 2019 Mar/Apr;39(2):267-277. doi: 10.11607/prd.3741. PMID 30794264
- [Background] Zuhr O, Baumer D, Hurzeler M. The addition of soft tissue replacement grafts in plastic periodontal and implant surgery: critical elements in design and execution. J Clin Periodontol. 2014 Apr;41 Suppl 15:S123-42. doi: 10.1111/jcpe.12185. PMID 24640997
- [Background] Wyrebek B, Gorski B, Gorska R. Patient morbidity at the palatal donor site depending on gingival graft dimension. Dent Med Probl. 2018 Apr-Jun;55(2):153-159. doi: 10.17219/dmp/91406. PMID 30152618
- [Background] Tseng ES, Tavelli L, Wang HL. Palatal Pedicle Flaps for Soft Tissue Augmentation. Int J Periodontics Restorative Dent. 2020 Jul/Aug;40(4):581-588. doi: 10.11607/prd.4561. PMID 32559041